CLINICAL TRIAL: NCT01275378
Title: COMPARATIVE EFFECTIVENESS RESEARCH FOR TWO MEDICAL HOME MODELS FOR ATTENTION DEFICIT HYPERACTIVITY DISORDER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Codman Square Health Center (Unknown); Dorchester House Health Center (Unknown)
Responsible Party: Principal Investigator, Michael Silverstein, Associate Professor of Pediatrics, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: R40MC17181
Record Dates: First submitted 2010-10-11; First posted 2011-01-12 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Care Plus (Active Comparator): Collaborative care model with specific theory-based elements to address common reasons for ADHD treatment failure
  Interventions: Behavioral: Collaborative Care Plus
- Traditional Collaborative Care (Active Comparator): Traditional collaborative care, in which care managers serve as intermediaries between primary care physicians and specialists
  Interventions: Behavioral: Traditional Collaborative Care

INTERVENTIONS:
Behavioral: Collaborative Care Plus — Traditional collaborative care + systematic addressing of ADHD comorbidities, parental mental health issues, and adherence to treatment plans
  Arms: Collaborative Care Plus
Behavioral: Traditional Collaborative Care — Traditional collaborative care, in which care managers serve as intermediaries between primary care physicians and specialists
  Arms: Traditional Collaborative Care

SUMMARY:
The purpose of this study is to compare the effectiveness of two care models on ADHD outcomes: one, a model of basic care management and structured communication with specialists, consistent with conventional descriptions of a patient-centered Medical Home; and another, which combines the Medical Home with theory-based care management strategies to address common reasons for ADHD treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Child is being evaluated for a potential diagnosis of ADHD by a primary care pediatrician at one of our sites.
* Child is 6 to 12 years of age
* Family plans to remain in the Boston area for the duration of the follow-up period
* Mother is comfortable in English or Spanish

Exclusion Criteria:

* Child already has a confirmed diagnosis of ADHD
* Child already receives ongoing specialty care in one or more of the following clinics: pediatric psychiatry, developmental behavioral pediatrics

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
ADHD Symptoms | 6 mo
  Swanson, Nolan and Pelham scale (SNAP-IV)
ADHD Symptoms | 12 mo
  Swanson, Nolan and Pelham scale (SNAP-IV)
Patient Medication Adherence | 6 mo
  Timely prescribed refills of ADHD medications - assessed through the EHR - will provide an accurate picture of medication adherence from the perspective of prescription writing. In addition, we will administer the validated Medication Adherence Scale, which has good reliability among parents of urban children with asthma
Patient Medication Adherence | 12 mo
  Timely prescribed refills of ADHD medications - assessed through the EHR - will provide an accurate picture of medication adherence from the perspective of prescription writing. In addition, we will administer the validated Medication Adherence Scale, which has good reliability among parents of urban children with asthma

SECONDARY OUTCOMES:
ODD Symptoms | 6 mo
  SNAP-IV
Social Skills | 6 mo
  Social Skills Rating System
Time to Symptom Improvement | 12 mo
  Based on follow-up ADHD symptom scales administered at regular intervals by our care managers, we will quantify the time between initial diagnosis and definitive improvement - conventionally defined by a 25% symptom reduction from baseline
ODD Symptoms | 12 mo
  SNAP-IV
Social Skills | 12 mo
  Social Skills Rating System

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Silverstein M, Hironaka LK, Walter HJ, Feinberg E, Sandler J, Pellicer M, Chen N, Cabral H. Collaborative care for children with ADHD symptoms: a randomized comparative effectiveness trial. Pediatrics. 2015 Apr;135(4):e858-67. doi: 10.1542/peds.2014-3221. PMID 25802346